CLINICAL TRIAL: NCT03576612
Title: Phase I Study of Neoadjuvant GMCI Plus Immune Checkpoint Inhibitor Combined With Standard of Care for Newly Diagnosed High-Grade Gliomas
Brief Title: GMCI, Nivolumab, and Radiation Therapy in Treating Patients With Newly Diagnosed High-Grade Gliomas
Acronym: GMCI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Candel Therapeutics, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABTC-1603; IRB00172749 (Other: JHM IRB); UM1CA137443 (NIH)
Record Dates: First submitted 2018-05-24; First posted 2018-07-03 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Glioma, Malignant
Keywords: glioblastoma, newly diagnosed, GMCI, Checkpoint inhibitor
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — Valacyclovir; Radiation; Radiotherapy; Temozolomide; Nivolumab

STUDY DESIGN:
Intervention Model Description: Newly diagnosed HGG: surgically eligible patients AdV-tk into wall of resection cavity; 1-3 days post-surgery Valacyclovir d1-14; Day 8 RT for 6 wks; day 15 TMZ 75mg/m2 daily; Nivo 240mgIV every 2 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: MGMT Unmethylated Patients (Experimental): After confirmation of high grade glioma, AdV-tk injection into wall of resection cavity. Valacyclovir starting 1-3 days post-surgery for 14 days. Radiation begins approximately day 8 and continues for 6 weeks. Temozolomide started after complete valacyclovir and stop when MGMT unmethylated result obtained. Nivolumab every 2 weeks x 26 doses up to 52 weeks. MRI every 8 weeks until progression.
  Interventions: Biological: AdV-tk; Drug: Valacyclovir; Radiation: Radiation; Drug: Temozolomide; Biological: Nivolumab; Other: Laboratory Biomarker Analysis
- Cohort 2: MGMT Methylated & undetermined Patients (Experimental): After confirmation of high grade glioma, AdV-tk injection into wall of resection cavity. Valacyclovir starting 1-3 days post-surgery for 14 days. Radiation begins approximately day 8. Temozolomide started after complete valacyclovir and continue during radiation then 5 week break and then begin adjuvant temozolomide dosing. Nivolumab every 2 weeks x 26 doses up to 52 weeks. MRI every 8 weeks until progression.
  Interventions: Biological: AdV-tk; Drug: Valacyclovir; Radiation: Radiation; Drug: Temozolomide; Biological: Nivolumab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: AdV-tk — Given IT
  Other Names: Aglatimagene Besadenovec
Drug: Valacyclovir — Given PO days 1-14; 1-3 days post surgery
  Other Names: 124832-26-4; L-Valine ester with 9-((2-hydroxyethoxy)methyl)guanine; Zelitrex
Radiation: Radiation — Undergo RT, 60Gy in 30 daily fractions M-F for 6weeks
  Other Names: Irradiate; irradiation; radiotherapy; RT
Drug: Temozolomide — Given PO during RT 75mg/m2 daily during RT Post RT cycle 1: 150mg/m2 days 1-5 150mg/m2 cycle 2-6: days 1-5 (150-200mg/m2)
  Other Names: TMZ
Biological: Nivolumab — day 15 post surgery 240mg IV q2wks x 26 doses , up to 52 weeks
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Other: Laboratory Biomarker Analysis — correlative studies

SUMMARY:
The purpose of this phase I trial is to test the safety of combining GMCI, an immunostimulator, plus nivolumab, an immune checkpoint inhibitor (ICI), with standard of care radiation therapy, and temozolomide in treating patients with newly diagnosed high-grade gliomas.

Gene Mediated Cytotoxic Immunotherapy (GMCI) involves the use of aglatimagene besadenovec (AdV-tk) injection into the tumor site and oral valacyclovir to kill tumor cells and stimulate the immune system. Nivolumab is an immune checkpoint inhibitor that may also stimulate the immune system by blocking the PD-1 immune suppressive pathway. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors and temozolomide is a chemotherapy drug that kills tumor cells. Giving GMCI, nivolumab, radiation therapy, and temozolomide may work better in treating patients with high-grade gliomas

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety/maximum tolerated dose (MTD) of the combination of aglatimagene besadenovec (AdV-tk) given intra-cranially at the time of initial tumor resection followed by valacyclovir (GMCI), nivolumab, and standard of care (radiation therapy [RT]+temozolomide [TMZ]) in patients with high-grade gliomas (HGG).

PRIMARY OBJECTIVES:

I. To assess the safety/maximum tolerated dose (MTD) of the combination of aglatimagene besadenovec (AdV-tk) given intra-cranially at the time of initial tumor resection followed by valacyclovir (GMCI), nivolumab, and standard of care (radiation therapy [RT]+temozolomide [TMZ]) in patients with high-grade gliomas (HGG).

SECONDARY OBJECTIVES:

I. To evaluate safety and toxicity of this combined treatment regimen. II. To estimate overall survival. III. To estimate progression free survival. IV. Immune biomarkers, including serum extracellular vesicles (EVs).

OUTLINE:

Patients undergo tumor resection and receive AdV-tk injection into the wall of the resection cavity. Patients then receive valacyclovir orally three times per day for 14 days. Beginning on approximately day 8, patients undergo radiation therapy five days per week for 6 weeks. Temozolomide will be initiated on approximately day 15 after valacyclovir is completed and will continue until MGMT methylation status is known. If unmethylated, temozolomide will be discontinued: these patients will constitute Cohort 1. In Cohort 2 - patients with methylated MGMT - temozolomide will continue. If methylation status is unable to be determined, those patients will also continue receiving temozolomide (Cohort 2). Both cohorts will receive nivolumab intravenously every two weeks for up to 52 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months for 2 years, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have operable brain tumor presumed to be high grade glioma (HGG) based on clinical and radiologic evaluation, where a gross total surgical resection of the contrast-enhancing area is intended; pathologic confirmation of HGG must be made at the time of surgery prior to AdV-tk injection, if not previously determined
* Patients must have a Karnofsky performance status >= 70% (i.e. the patient must be able to care for himself/herself with occasional help from others)
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Hemoglobin >= 9 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN), (except for patients with known Gilbert's syndrome who must have normal direct bilirubin)
* Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransaminase (ALT) serum glutamate pyruvate transaminase (SGPT) =< 3.0 x institutional ULN
* Creatinine =< institutional ULN
* Calculated creatinine clearance >= 40 ml/min (use a modified Cockcroft-Gault equation)
* Activated partial thromboplastin time/partial thromboplastin time (APTT/PTT) =< 1.5 x institutional ULN
* Patients must be able to provide written informed consent
* Patients must have magnetic resonance imaging (MRI) within 14 days of starting treatment; patients must be able to tolerate MRI
* Women of childbearing potential must agree to have a negative serum pregnancy test within 24 hours prior to treatment start; women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study treatment, and through at least 5 months after the last dose of study drug; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; sexually active men of reproductive potential who are partners of women with reproductive potential must also agree to use adequate contraception prior to the study, for the duration of study participation, and through at least 7 months after the last dose of study drug; adequate methods of effective birth control include sexual abstinence (men, women); vasectomy; or a condom with spermicide (men) in combination with barrier methods, hormonal birth control or intrauterine device (IUD) (women)
* Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder; patients with prior malignancies must be disease-free for >= two years; patients with low-risk prostate cancer on active surveillance are eligible
* Patients must be able to swallow oral medications
* Patients must not have received prior radiation therapy, chemotherapy, immunotherapy or therapy with biologic agent (including immunotoxins, immunoconjugates, antisense, peptide receptor antagonists, interferons, interleukins, tumor infiltrating lymphocyte [TIL], lymphokine-activated killer [LAK] or gene therapy), or hormonal therapy for their brain tumor; glucocorticoid therapy is allowed

Exclusion Criteria:

* Patients receiving any other investigational agents are ineligible
* Patients with a history of hypersensitivity or allergic reactions attributed to compounds of similar chemical or biologic composition to valacyclovir, acyclovir, or temozolomide are ineligible; the valacyclovir and temozolomide package inserts can be referenced for more information
* Patients with a history of severe hypersensitivity reaction to any monoclonal antibody are ineligible
* Patients who require therapy with systemic immunosuppressive drugs except corticosteroids are ineligible
* Patients with a history of active autoimmune disease requiring treatment in the past 2 years are ineligible
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active liver disease or active hepatitis, or psychiatric illness/social situations that would limit compliance with study requirements, are ineligible
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with these agents through 1 week after receiving the last dose of study drugs
* Patients who are known to be human immunodeficiency virus (HIV) positive are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 2 years
  National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 will be used for scoring toxicity and adverse events. The severity and frequency of toxicity will be tabulated by the tested dose or doses using descriptive statistics. The proportions of subjects who experienced grade 3 or above toxicities will be estimated, along with 95% confidence intervals by each type of toxicity.

SECONDARY OUTCOMES:
Overall survival (death) | From initial diagnosis to the date of death/or censored at the time of last known alive, assessed for up to 2 years
  To estimate overall survival - endpoint is death. Median time of survival along with 95% confidence interval will be estimated using the Kaplan-Meier method.
Progression-free survival (progression) | From initial diagnosis to the date progression is defined, assessed for up to 2 years
  To estimate progression-free survival - endpoint is progression. Median time of progression-free survival along with 95% confidence interval will be estimated using Kaplan-Meier method.
Immune profiling - Tumor Tissue | Up to 2 years
  Tumor profiling by immunohistochemistry and Nanostring at baseline and when samples available after treatment.
Tumor mutation - Tumor Tissue | Up to 2 years
  Mutational profiling by sequence or transcriptome analysis from tumor tissue
Peripheral blood mononuclear cells (PBMCs) in serum samples | Up to 2 years
  Standard descriptive statistics will be used to summarize proportion of PBMCs.
Immune characterization as determined by Cytokines | Up to 2 years
  Immune characterization of surface and content proteins is determined by presence of cytokines in serum.
Immune characterization as determined by Extracellular vesicles (EVs) proteins | Up to 2 years
  Immune characterization of surface and content proteins based on presence of extracellular vesicles in serum samples.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wen, MD, Study Chair — Dana Farber
Locations (5):
- United States (5):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Abrams Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wen PY, Manzanera A, Duault C, Gonzalez-Kozlova E, Lopez L, Grossman SA, Ye X, Fisher J, Lee I, Walbert T, Snyder J, Brem S, Desai A, Bagley SJ, Kakani C, Strowd R, Tatter S, Laxton A, Lesser G, Amankulor N, Lieberman F, Drappatz J, Mantica M, Triggs D, Haymaker C, Wistuba II, Al-Atrash G, Mendoza Perez J, Futreal A, Little LD, Islam MDH, Duose D, Jiang P, Reuben A, Lawler SE, Pichavant M, Gentles A, Bendall S, Kong A, Camacho C, Del Valle D, Kim-Schulze S, Gnjatic S, Sharon E, Nowicki MO, Peruzzi P, Lane D, Aguilar-Cordova E, Aguilar LK, Nichols G, Dwyer J, Tak PP, Maecker H, Barone F, Chiocca EA. A multi-institutional phase 1 clinical trial exploring upfront multimodal standard of care and combined immunotherapies for newly diagnosed glioblastoma. Neuro Oncol. 2025 Mar 22:noaf079. doi: 10.1093/neuonc/noaf079. Online ahead of print. PMID 40120123